CLINICAL TRIAL: NCT00890409
Title: Selective Head Cooling With Mild Systemic Hypothermia After Neonatal Hypoxic-Ischemic Encephalopathy: A Multi-Center Randomized Controlled Trial in China
Brief Title: Safety and Efficacy of Hypothermia to Treat Neonatal Hypoxic-Ischemic Encephalopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Qingdao Children's Hospital (Unknown); Guangxi Maternity and Infant health Hospital (Unknown); Quanzhou Children's Hospital (Other); The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Xiaomei Shao, Children's Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Engineering 211
Record Dates: First submitted 2009-01-02; First posted 2009-04-29 (Estimated); Results first posted 2009-04-29 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: hypothermia; neonate; hypoxic-ischemic encephalopathy; efficacy; safety
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normothermia (No Intervention): Rectal temperature was maintained at 36.0-37.5 degree C.
- Hypothermia (Experimental): The group was fitted with a cooling cap around the head for 72 hours. The temperature of the cap could be adjusted between 5 to 20 degree C and was automatically regulated by a servo-controlled temperature probe placed in the nasopharynx to maintain the nasopharyngeal temperature at (34±0.2)degree C. All infants were nursed under a servo-controlled radiant warmer and the rectal temperature was maintained at 34.5 to 35 degree C. Head cooling was started within 6 hours after birth for 72 hours followed by spontaneous re-warming and the average time to reach the target temperature was 2 hours.
  Interventions: Device: Cooling cap (YJW608-04B)

INTERVENTIONS:
Device: Cooling cap (YJW608-04B) — A semiconductor water circulation cooling device (YJW608-04B, Henyang Radio Manufactory, Hunan, China) was used to conduct head cooling. The hypothermia group was fitted with a cooling cap around the head for 72 hours. The temperature of the cap could be adjusted between 5 to 20 degree C and was automatically regulated by a servo-controlled temperature probe placed in the nasopharynx to maintain the nasopharyngeal temperature at (34±0.2)degree C. All infants were nursed under a servo-controlled radiant warmer and the rectal temperature was maintained at 34.5 to 35 degree C. Head cooling was started within 6 hours after birth for 72 hours followed by spontaneous re-warming and the average time to reach the target temperature was 2 hours.
  Other Names: YJW608-04B
  Arms: Hypothermia

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of selective head cooling (SHC) in neonatal hypoxic-ischemic encephalopathy (HIE).

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) remains a major cause of neonatal death and long term disabilities. Data from animal studies have shown protective effects of mild hypothermia to both the mature and immature brain. Recently research priorities have moved from bench to bedside. Several studies have shown a trend for brain protection of mild to moderate hypothermia and mild hypothermia has emerged as a promising treatment for HIE. Therefore,the investigators organized a multi-centered randomized controlled trial of selective head cooling (SHC) combined with mild systemic hypothermia in HIE newborn infants.

ELIGIBILITY:
Inclusion Criteria:

* Age up to 6 hours
* Gestational age ≥ 36 weeks and birth weight ≥ 2500 g
* Apgar score ≤ 3 at 1 minute and ≤ 5 at 5 minutes, and/or cord blood gas pH < 7.0 or base deficit ≤ 16 mmol/L, and/or need for resuscitation or ventilation at 5 minutes of age
* Clinical signs of encephalopathy (seizures, coma, abnormal muscle tone and irregular breathing, etc)

Exclusion Criteria:

* Major congenital abnormalities
* Infection
* Other etiology of induced brain injury
* Severe anemia (Hb < 120 g/L)

Eligible infants assessed for the severity of HIE according to criteria of the Neonatal Association of Chinese Academy of Pediatrics 25 modified from Sarnat and Sarnat 26 in 1986

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2002-05; Primary Completion 2004-06 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, M.D, Study Chair — Children's Hospital, Fudan University
Locations (1):
- Children's Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Gluckman PD, Wyatt JS, Azzopardi D, Ballard R, Edwards AD, Ferriero DM, Polin RA, Robertson CM, Thoresen M, Whitelaw A, Gunn AJ. Selective head cooling with mild systemic hypothermia after neonatal encephalopathy: multicentre randomised trial. Lancet. 2005 Feb 19-25;365(9460):663-70. doi: 10.1016/S0140-6736(05)17946-X. PMID 15721471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: May 2002 to August 2005; Types of location: Children's Hospital or Women and Children's Medical Centre.
Groups:
- Normothermia: Rectal temperature in the group was maintained at 36 to 37.5 degree C.
- Hypothermia: The group was fitted with a cooling cap around the head for 72 hours. The temperature of the cap could be adjusted between 5 to 20 degree C and was automatically regulated by a servo-controlled temperature probe placed in the nasopharynx to maintain the nasopharyngeal temperature at (34±0.2)degree C.
Period: Overall Study
Arm/Group | Normothermia | Hypothermia
Started | 116 | 140
Completed | 96 | 119
Not Completed | 20 | 21
Not completed — Lost to Follow-up | 20 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normothermia | Hypothermia | Total
Number analyzed (Participants) | 116 | 140 | 256
Age, Customized [Mean (Standard Deviation); unit: hour]
  <=6 hours | 4.03 (1.21) | 4.12 (1.59) | 4.07 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 97 | 115 | 212

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: The number of deaths by 18 months of age.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 96 | 119
participants | 27 | 22

2. Primary Outcome: Severe Neurodevelopmental Disability
Description: Severe disability was defined as cerebral palsy (CP) or mental retardation (MR). The definition of MR was development quotient (DQ) <70 by Gesell's Child Development Scale and CP was based on the Criteria of a level 3 to 5 by the Gross Motor Function Classification System (GMFCS).
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 69 | 97
participants | 19 | 11

3. Secondary Outcome: Major Adverse Events
Description: Major adverse events were defined as severe arrhythmia (II or III degree A-V block or atrial or ventricular arrhythmia), major venous thrombosis, refractory hypotension (mean blood pressure less than 40 mmHg), moderate or severe scleredema (greater or equal to 20% body surface area), and severe bleeding.
Time Frame: 18 months
Measure: Number; unit: participants
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 96 | 119
participants | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No